CLINICAL TRIAL: NCT07081763
Title: Immunotherapy With a JAK1/JAK2 Inhibitor (Baricitinib) and an mTORC1 Inhibitor (Sirolimus), Alone and in Combination, for the Control of HIV-1 Replication After Antiretroviral Treatment Interruption: a Phase II Multicenter, Multi-arm, Multi-stage, Randomized, Double-blind, Placebo-controlled, Adaptative Trial
Brief Title: Immunotherapy With Baricitinib and Sirolimus, Alone and in Combination, for the Control of HIV-1 Replication After Antiretroviral Treatment Interruption
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANRS 0668s RHIVIERA-03; 2025-523118-97-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-11; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
Keywords: Antiretroviral Treatment Interruption
MeSH Terms: interventions — baricitinib; Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- baricitinib + placebo of sirolimus (Experimental): baricitinib : participants will receive a 10-week course of baricitinib from W0 to W10, starting 2 weeks before the ATI period (ARV stop at W2) and ending 8 weeks after (W10). Baricitinib will be administered orally at 2 mg QD from W0 to W10.
  placebo of sirolimus : participants will receive a 10-week course of sirolimus placebo from W0 to W10, starting 2 weeks before the ATI period (starting at W2) and ending 8 weeks after (W10).
  Interventions: Drug: Baricitinib 2 MG; Other: Placebo of sirolimus 2 MG
- sirolimus + placebo of baricitinib (Experimental): sirolimus : participants will receive a 10-week course of sirolimus from W0 to W10, starting 2 weeks before the ATI period (ARV stop at W2) and ending 8 weeks after (W10). Sirolimus will be administered orally at 2 mg QD.
  placebo of baricitinib : participants will receive a 10-week course of baricitinib placebo from W0 to W10, starting 2 weeks before the ATI period (starting at W2) and ending 8 weeks after (W10).
  Interventions: Drug: Sirolimus 2 MG; Other: Placebo of baricitinib 2 MG
- baricitinib + sirolimus (Experimental): baricitinib : participants will receive a 10-week course of baricitinib from W0 to W10, starting 2 weeks before the ATI period (ARV stop at W2) and ending 8 weeks after (W10). Baricitinib will be administered orally at 2 mg QD from W0 to W10.
  sirolimus : participants will also receive a 10-week course of sirolimus from W0 to W10, starting 2 weeks before the ATI period (ARV stop at W2) and ending 8 weeks after (W10). Sirolimus will be administered orally at 2 mg QD.
  Interventions: Drug: Baricitinib 2 MG; Drug: Sirolimus 2 MG
- placebo of baricitinib + placebo of sirolimus (Placebo Comparator): Participants will receive a 10-week course of both baricitinib placebo and sirolimus placebo from W0 to W10, starting 2 weeks before the ATI period (starting at W2) and ending 8 weeks after (W10).
  Interventions: Other: Placebo of baricitinib 2 MG; Other: Placebo of sirolimus 2 MG

INTERVENTIONS:
Drug: Baricitinib 2 MG — Administered orally at 2 mg QD from W0 to W10.
  Arms: baricitinib + placebo of sirolimus; baricitinib + sirolimus
Drug: Sirolimus 2 MG — Administered orally at 2 mg QD from W0 to W10.
  Arms: baricitinib + sirolimus; sirolimus + placebo of baricitinib
Other: Placebo of baricitinib 2 MG — Administered orally at 2 mg QD from W0 to W10.
  Arms: placebo of baricitinib + placebo of sirolimus; sirolimus + placebo of baricitinib
Other: Placebo of sirolimus 2 MG — Administered orally at 2 mg QD from W0 to W10.
  Arms: baricitinib + placebo of sirolimus; placebo of baricitinib + placebo of sirolimus

SUMMARY:
Natural HIV controllers (HICs) and post-treatment controllers (PTCs) are rare examples of people living with HIV (PLWH) who achieve control of HIV replication without the need for antiretroviral therapy (ART). Therapeutic strategies that can induce such a phenotype are therefore a key goal in the quest for a remission of HIV infection.

JAK1/JAK2 and mTORC1 are key biological pathways involved in the regulation of HIV-1 transcription and replication, as well as the functional capacities of immune effectors, primarily CD8 T cells (exhaustion status and immunometabolic properties), but also NK cells. Immunotherapeutic interventions using a JAK1/JAK2 inhibitor and an mTORC1 inhibitor, alone or in combination to achieve an additive or synergistic effect, are therefore promising candidates to induce a PTC-like phenotype. The use of combined approaches of immunotherapies with different and potentially complementary effects may increase the likelihood of achieving viral control.

This study aims at evaluating the efficacy and safety of three experimental immunotherapeutic interventions (i.e., baricitinib, a JAK1/JAK2 inhibitor, alone; sirolimus, an mTORC1 inhibitor, alone; or their combination) on viral control following an analytic treatment interruption (ATI) of antiretroviral drugs in PLWH who had initiated ART during primary HIV-1 infection. This randomized clinical trial will use an innovative multi-arm multi-stage adaptive design.

DETAILED DESCRIPTION:
This phase II multicenter, multi-stage, randomized, double-blind, placebo-controlled, adaptive clinical trial will evaluate the effect of baricitinib and sirolimus, alone and in combination, on viral control following an analytical treatment intervention (ATI).

The trial will follow an adaptive multi-arm multi-stage (MAMS) design. It will be divided into three stages, two interim stages and one final stage. Recruitment in any arm may be stopped early if, in the opinion of the Independent Data Monitoring Committee (IDMC), an experimental arm is considered to have insufficient efficacy or for safety reasons. The final sample size and study duration will depend on how many arms are continued beyond the interim analyses

Participants will be randomized 1:1:1:1 to either one of 4 arms:

* Arm 1: baricitinib + placebo of sirolimus
* Arm 2: sirolimus + placebo of baricitinib
* Arm 3: baricitinib + sirolimus
* Arm 4: placebo of baricitinib + placebo of sirolimus

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years and ≥ 65 years,
* Weight ≥ 50 kg and ≤ 100 kg,
* HIV-1 infection having been diagnosed at primary infection stage with an HIV-1 RNA VL > 1,000 copies/mL and either a negative or incomplete WB [0-5] bands or IB [0-3] bands and/or a previous negative HIV-1 ELISA within the past 3 months,
* Having initiated ART within 2 months of primary HIV-1 infection diagnosis,
* Having received ART continuously without interruption,
* Receiving ART for at least 1 year prior to enrollment,
* Receiving DTG-, BIC-, RAL-, or RPV-based ART (PI-, EVG/c-, NVP-, EFV-, ETR- or DOR-based ART must have been switched to DTG-, BIC-, RAL-, or RPV-based ART at W-8).
* Sustained HIV-1 plasma viral load ≤ 50 copies/mL for ≥ 6 months prior to enrollment (with at least two measurements, including the screening value),
* Blood CD4 T-cell count ≥ 500 cells/µL (on the last two measurements, including screening),
* Willing to interrupt ART for ATI and change ART regimen before if required to avoid drug-drug interactions,
* Willing to take valaciclovir 500 mg QD from W0 to W10 to prevent recurrence of herpes or herpes zoster,
* If sexually active, willing to use a reliable method of reducing the risk of transmission to their sexual partners during treatment interruption (condoms or PrEP for their sexual partners).
* If able to have children, willing to use a highly effective method of contraception (combined oral contraceptive pill; implanted contraceptive device, IUD/IUS; physiological or anatomical sterility for self of partner); willing to undergo blood bHCG at screening and before ATI.
* Willing to comply with visit schedule and provide blood samples according to the protocol.
* Written informed consent (at the latest on the day of the enrollment visit and before any exams to be performed in the context of the trial) (article L1122-1-1 of the French CSP).
* Participant covered by Health Insurance (article L1121-11 of the French CSP).

Exclusion Criteria:

* HIV-2 infection,
* Previous interruption of ART,
* Loss of virologic suppression (VL > 200 c/mL) at any time while on effective ART; previous blips of VL between 50 and 200 c/mL allowed, except in the 6 months prior to screening,
* Long-acting ART based on CAB/RPV, lenacapavir, islatravir, or ibalizumab,
* Receiving PI-, EVG/c-, NVP-, EFV-, ETR- or DOR-based ART beyond W-8,
* No other active ARV regimen in addition to the current one,
* Pregnant or lactating woman,
* Woman expecting to conceive during the trial period,
* Any medical condition that will contraindicate an interruption of ARV treatment,
* History of coronary artery disease, stroke, or blood clots; thrombophilia,
* High cardiovascular risk (SCORE2 ≥ 7.5% if < 50 years, or ≥ 10% if 50-65 years),
* Active cancer or history of cancer,
* Active opportunistic infection,
* Active or latent tuberculosis (unless prophylaxis has been received in the past); participant must be screened for latent tuberculosis according to routine practice prior to initiation of immunotherapeutic interventions,
* Chronic hepatitis B (positive HBs antigen and/or positive HBV DNA) or past-hepatitis B infection (positive anti-HBc antibodies) or hepatitis C (positive HCV RNA); cirrhosis,
* Treatment with systemic corticosteroids or immunosuppressants currently or within 12 weeks prior to study randomization,
* History of experimental vaccination against HIV,
* Ongoing treatment with strong CYP3A4 inducers or inhibitors,
* History of hypersensitivity to macrolides.

Laboratory parameters at screening:

* Polynuclear neutrophils <1 G/L; Hemoglobin <10 g/dL; Platelets <100 G/L
* GFR <30 ml/min/1.73m2
* TP <50%; ALAT/ASAT >5x ULN; Bilirubin >3x ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the time to restart of ART due to virological rebound or a clinical decision to restart ART due to CD4 T-cell decline, an AE, or for any other reason | 26 weeks